CLINICAL TRIAL: NCT00921908
Title: Multihole or Epidural Catheter for Local Anesthetic in the Wound
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Other Study IDs: H-A-2008-028
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Postoperative Pain; Hip Arthroplasty
Keywords: total hip arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Sodium Chloride

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- epidural catheter: subfascial placement of a triple-orifice epidural catheter
  Interventions: Other: 2 mBq radioactive technetium diluted in 20 mL saline
- multiholed catheter: subfascial placement of a multi-orifice 15 cm catheter
  Interventions: Other: 2 mBq radioactive technetium diluted in 20 mL saline

INTERVENTIONS:
Other: 2 mBq radioactive technetium diluted in 20 mL saline

SUMMARY:
Postoperative administration of local anesthetics is effective for postoperative pain management across surgical specialties but the optimal type of catheter (single, few or multiholed catheters) has not been determined.

This study investigates wound spread of a radioactive isotope (technetium) administered in different types of catheters after total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* operation with total hip arthroplasty

Exclusion Criteria:

* allergies to drugs administered

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients undergoing total hip arthoplasty
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
wound spread area of radioactive isotope

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark